CLINICAL TRIAL: NCT05047094
Title: A Safety and Efficacy Study of Intratumoral Diffusing Alpha Radiation Emitters in Recurrent Unresectable or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Safety and Efficacy Study for Combinational Treatment of DaRT and Check Point Inhibitor for Recurrent Unresectable or mHNSCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-HNCPI-00
Record Dates: First submitted 2021-08-29; First posted 2021-09-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Skin Cancer; Metastatic Head-and-neck Squamous-cell Carcinoma
Keywords: Squamous Cell Carcinoma; SCC; Skin Cancer; Skin metastasis; HNSCC; Carcinoma, Squamous; Recurrent disease; Alpha radiation; Brachytherapy; Pembrolizumab; Check Point Inhibitor; KEYTRUDA; Immunomodulators
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Skin Neoplasms; Carcinoma, Squamous Cell; Recurrence | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DaRT seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds in Combination with Standard Treatment of Pembrolizumab
  Interventions: Device: Diffusing Alpha Radiation Emitters Therapy (DaRT); Drug: Pembrolizumab

INTERVENTIONS:
Device: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms.
  Other Names: DaRT
Drug: Pembrolizumab — 200 mg administered as an intravenous infusion over 30 minutes every 3 weeks
  Other Names: KEYTRUDA

SUMMARY:
A unique combinational treatment for cancer employing intratumoral diffusing alpha radiation emitter device with check point inhibitor for recurrent unresectable or metastatic Head and Neck Squamous Cell Carcinoma

DETAILED DESCRIPTION:
This will be a prospective, open-label, one arm, single center two-stage adaptive trial designed to stop for either futility or efficacy after the first stage.

This approach will combine Diffusing Alpha Radiation Emitters seeds implantation along with standard treatment of Pembrolizumab for patients with recurrent unresectable or metastatic Head and Neck Squamous Cell Carcinoma (mHNSCC).

The DaRT seeds will be implanted in the target lesion and removed 15-22 days after implantation. Concurrently, patient will receive standard treatment of Pembrolizumab.

Disease evaluation will be assessed by a radiological imaging every 6 weeks starting at day 42 after the DaRT insertion procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed, metastatic, or recurrent unresectable squamous cell carcinoma of the head and neck.
2. Ability to provide tissue sample, either from an archive or undergo another biopsy to provide a fresh sample
3. Targetable lesion must be technically amenable for the DaRT seeds implantation
4. Brachytherapy indication validated by a multidisciplinary team
5. Targetable lesion according to RECIST v1.1
6. Age ≥ 18 years old
7. Eastern Cooperative Oncology Group (ECOG) Performance Status Scale ≤ 2
8. Subjects' life expectancy is more than 6 months
9. White Blood Count (WBC) ≥ 3500/µl, granulocyte ≥ 1500/µl
10. Platelet count ≥ 100,000/µl
11. Hemoglobin ≥ 9 g/dl
12. Calculated or measured creatinine clearance ≥ 60 cc/min
13. Aspartate Aminotransferase (AST) and Alanine Transaminase (ALT) ≤ 2.5 X Upper Limit of Normal (ULN) or ≤ 5 X ULN for subjects with liver metastases
14. International normalized ratio (INR) <1.4 for patients not on Warfarin
15. Subjects are willing and able to sign an informed consent form
16. Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test before the Ra-224 implantation and are required to use an acceptable contraceptive method to prevent pregnancy for 3 months after brachytherapy.

Exclusion Criteria:

1. Previous treatment for metastatic disease (for recurrent unresectable disease, previous treatment is allowed given that 6 months had elapsed from completion of treatment for primary disease)
2. Patients with brain metastases
3. Combined Positive Scores (CPS) <1
4. Patients with known contraindications to radiotherapy
5. Any prior therapy with anti-PD-L1 (Programmed death-ligand), anti-PD-L2, anti-CTLA-4 (Cytotoxic T lymphocyte antigen) antibody, etc.
6. Any history of a sever hypersensitivity reaction to any monoclonal antibody.
7. Known hypersensitivity to any of the components of the DaRT.
8. Has a known history of active TB (Tuberculosis Bacillus )
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
10. Any diagnosis of immunodeficiency or current immunosuppressive therapy including >10mg/day of prednisone within 14 days of enrollment is not permitted
11. Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
12. Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
13. Patient requires treatment which may conflict with the endpoints of this study including evaluation of response or toxicity of DaRT.
14. Has a known history of Human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
15. Has known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected)
16. Pregnancy or lactation.
17. Patients must agree to use adequate contraception (abstinence, barrier method of birth control, or any other medically acceptable form of contraception) prior to study entry, for the duration of study participation and for 6 months after last dose of Pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Efficacy of DaRT Treatment in Combination with Pembrolizumab | From Day 26 to date of documented best response, assessed up to 24 months
  Assessed via the Confirmed Best Overall Response (BOR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST Version 1.1)

SECONDARY OUTCOMES:
Adverse Events | Until completion of the last study-related procedure, approximately 2 years
  Assessment of the frequency, severity and causality of acute adverse events related to the DaRT treatment in combination with immune checkpoint inhibitors. This will be assessed and graded according to Common Terminology and Criteria for Adverse Events (CTCAE) version 5.0. (graded 1-5, 1 is mild and 5 is death)
Progression Free Survival (PFS) | From first dose of Pembrolizumab until progressive disease is recorded (up to 24 months)
  PFS will be defined as time from Pembrolizumab treatment start date to progressive disease according to RECIST v1.1 or death due to any cause, whichever occurs first
Overall Survival (OS) | From Pembrolizumab treatment start date to death or lost to follow-up (up to 24 months)
  Defined as the time from Pembrolizumab treatment start date to death due to any cause or lost to follow up.
Duration of Response (DOR) | From first record of response until the first date recurrent or progressive disease is documented (up to 24 months)
  Duration of response is defined as the interval from the time measurement criteria are first met for Complete Response (CR), Partial Response (PR), or Stable Disease (SD) (whichever is first recorded) until the first date recurrent or progressive disease is objectively documented.

OTHER OUTCOMES:
Change in Expression of Immune-Related Biomarkers | On Day -16, day 0, day 15, and day 68
  This study will assess the change in immune related biomarkers in peripheral blood using Fluorescence-activated cell sorting (FACS) analysis. These biomarkers include: CD3, CD4, CD8, CD69, CD137

CONTACTS AND LOCATIONS:
Overall Officials: Aron Popovtzer, MD, Principal Investigator — Sharett institute, Hadassah Medical Center - Ein-Kerem
Locations (3):
- Israel (3):
  - Sharett institute, Hadassah University Hospital - Ein-Kerem, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel-Aviv Medical Center, Tel Aviv